CLINICAL TRIAL: NCT04719091
Title: CLINICAL EVALUATION OF THE EFFICACY OF AN INTRA ORAL SPRAY FOR PATIENTS WITH XEROSTOMIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: You First Services (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LUX-101-15
Record Dates: First submitted 2021-01-20; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Dry Mouth, Xerostomia.Hyaluronic Acid, Xylitol
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Triple(Participant, Care provider, investigator)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HA formulation Oral Spray (Experimental): The Study Examiner and staff will screen for subjects that meet the enrollment criteria. Subjects will be randomly assigned to one of two treatment groups. Oral soft and hard tissue examinations will be conducted at each visit. Following an initial 3-5 minute evaluation of resting salivary flow, subjects will wait 10 minutes and then use their assigned spray. They will then swallow, and unstimulated saliva will be collected for 3-5 minutes. They will then remain in the study center for 60 min to evaluate xerostomia relief by questionnaire at 5, 15, 30, 45 and 60 min. after the use of Experimental mouth spray. They will then be given their assigned product to use twice daily for one week
  Interventions: Device: Lubricity
- Placebo Oral Spray (Placebo Comparator): The Study Examiner and staff will screen for subjects that meet the enrollment criteria. Subjects will be randomly assigned to one of two treatment groups. Oral soft and hard tissue examinations will be conducted at each visit. Following an initial 3-5 minute evaluation of resting salivary flow, subjects will wait 10 minutes and then use their assigned spray. They will then swallow, and unstimulated saliva will be collected for 3-5 minutes. They will then remain in the study center for 60 min to evaluate xerostomia relief by questionnaire at 5, 15, 30, 45 and 60 min. after the use of placebo mouth spray. They will then be given their assigned product to use twice daily for one week
  Interventions: Device: Lubricity

INTERVENTIONS:
Device: Lubricity — Oral spray

SUMMARY:
This cross-over group, double-blind, randomized, single center, study will enroll 26 subjects to target at least 24 subjects completing the study.Following an initial 3-5 minute evaluation of resting salivary flow, subjects will wait 10 minutes and then use their assigned spray. They will then swallow, and unstimulated saliva will be collected for 3-5 minutes. They will then remain in the study center for 60 min to evaluate xerostomia relief by questionnaire at 5, 15, 30, 45 and 60 min. after the use of mouth spray. They will then be given their assigned product to use twice daily for one week. Subjects will maintain a daily diary of their use of the mouth spray and any oral effects they experience, and will answer all diary questions. Compliance will be assessed by subject diary and measurement of remaining test mouth spray in bottle when unused portion is returned to the clinic. Subjects will also receive 2 questionnaires to complete during the office visit at the end of each 7-day study period. After a 1 week washout, subjects will return to the office to begin the second period of the study, using the same study procedures and be assigned the alternate treatment mouth spray.

ELIGIBILITY:
Inclusion Criteria:

* Have provided written informed consent prior to being entered into the study.
* Must be at least 18 years of age, male or female.
* Have at least 12 natural or restored teeth.
* Have a negative history of radiation therapy to head and neck
* Have a complaint of xerostomia
* Have an unstimulated salivary flow rate <0.25ml/minute which represents 35-50% of normal salivary function
* Agree not to have a dental prophylaxis or any other elective, non-emergency dental procedures (other than those provided during the study) any time during the study.
* Agree to abstain from the use of any products for xerostomia other than those provided in the study.
* Agree to comply with the conditions and schedule of the study.

Exclusion Criteria:

* Physical limitations or restrictions that might preclude normal tooth brushing.
* Evidence of gross oral pathology, including widespread caries or chronic neglect, extensive restoration, pre-existing gross plaque or soft or hard tissue tumor of the oral cavity.
* Presence of severe gingivitis with 30 or more sites showing bleeding on probing.
* Evidence of major oral hard or soft tissue lesions or trauma at the baseline visit as determined by the Investigator/Examiner.
* Chronic disease with concomitant oral manifestations other than xerostomia
* Conditions requiring antibiotic treatment prior to dental prophylaxis and invasive procedures, such as heart murmur, history of rheumatic fever, valvular disease or certain prosthetic implants.
* History of uncontrolled diabetes or hepatic or renal disease, or other serious conditions or transmittable diseases, (e.g. cardiovascular disease, AIDS).
* Subjects who are currently undergoing, or require, extensive dental work or orthodontic treatment.
* Currently using bleaching trays.
* History of significant adverse effects following use of oral hygiene products such as toothpastes and mouth sprays.
* Subjects who are nursing, pregnant or plan to become pregnant for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-01-02 (Actual); Primary Completion 2016-02-01 (Actual); Study Completion 2016-02-29 (Actual)

PRIMARY OUTCOMES:
Relief from dry mouth using VAS scoring | 3 weeks
  At end of each treatment week they will be asked to answer the following VAS question
  How well did this product make your mouth feel moist? At end of each treatment week they will be asked to answer the following VAS question
  At the end of the study they will be asked: How would you rate the second mouthspray compared to the first Study mouthspray in terms of your mouth feeling moist?